CLINICAL TRIAL: NCT05367024
Title: Broccoli Effect on Glycated Haemoglobin (HbA1c) - BETA Study, A Randomised Double-blinded Crossover Study
Brief Title: Broccoli Effect on Glycated Haemoglobin (HbA1c)
Acronym: BETA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: QIB06-2020
Record Dates: First submitted 2021-10-04; First posted 2022-05-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pre-diabetes
Keywords: Broccoli; Pre-diabetes; Glycated Haemoglobin (HbA1c); Glucose; Energy metabolism
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Broccoli soup (Experimental): The soup will be made with a commercially available dried vegetable soup supplemented with broccoli powder.
  Interventions: Other: Broccoli soup
- Courgette soup (Sham Comparator): The soup will be made with a commercially available dried vegetable soup supplemented with courgette powder.
  Interventions: Other: Courgette soup

INTERVENTIONS:
Other: Broccoli soup — Participants will consume one broccoli soup three times a week for one 12-week intervention period as part of their normal diet.
  Arms: Broccoli soup
Other: Courgette soup — Participants will consume one courgette soup three times a week for one 12-week intervention period as part of their normal diet.
  Arms: Courgette soup

SUMMARY:
Broccoli has shown to normalise elevated blood sugars when eaten over long period of time. Individuals with pre-diabetes have higher than normal blood sugar levels. In this study, investigators are trying to understand how broccoli, when eaten as a soup, affects blood sugar levels in individuals with pre-diabetes.

DETAILED DESCRIPTION:
The BETA study is a 36-week randomized, double-blind, placebo-controlled, two-arm crossover intervention study conducted at the Quadram Institute Clinical Research Facility (QI CRF), Norwich, UK. Investigators are seeking adults with pre-diabetes, to determine whether broccoli soups affect glucose metabolism, compared to a similar soup containing courgette. There are a total of 9 clinical visits (1 screening visit, 4 short visits, and 4 oral glucose tolerance testing visits). Investigators will assess blood samples for glycated hemoglobin (HbA1c), fasting plasma glucose, insulin, fructosamine, cholesterol and triglycerides. Investigators will also quantify the metabolites in urine through analytical analysis and determine whether gene expression is altered by the soups through RNA sequencing. Participants will consume one of two soups (broccoli or courgette) for the first intervention period then after a twelve-week washout phase (soup holiday), participants will crossover and consume the other soup for the second intervention period. For each intervention period, soups will be consumed three times a week per twelve-week period. Investigators will ask the participant to complete lifestyle questionnaires regarding their physical activity and dietary pattern.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with prediabetes (confirmed through screening)
* Aged 18 and older.
* Body Mass Index (BMI) between 18.5 - 35 kg/m2.
* Living within 40 miles from the Norwich Research Park.

Exclusion Criteria:

The participant will not be able to take part if they('re):

* Screening test results indicate they are not suitable to take part in this study such as HbA1c level at screening visit of < 42 mmol/mol (healthy) and > 47 mmol/mol (diabetes) and BMI at screening visit < 18.5 kg/m2 (underweight) and > 35 kg/m2 (extremely obese).
* Have a known allergy to any of the components (broccoli, courgette, milk, lactose, or gluten) of the test soups.
* Have been diagnosed or have a history of blood or clotting disorders such as anaemia or thrombosis.
* Have been treated for heart disease, cancer, or diabetes.
* Are immunocompromised due to medications or viral infection such human immunodeficiency virus (HIV).
* Have low or high blood pressure with hypertension medication (≤90/60, ≥160/100 respectively would be classed as abnormal).
* Have any acute or chronic illnesses that affects the outcome of the study such as a gastrointestinal disorder. This will be assessed on a case by case basis by QI medical advisor.
* Plan to become pregnant during the study duration, pregnant or breastfeeding.
* Frequently take medications that may interfere with sugar metabolism or absorption such as laxatives, steroids, dietary supplements, or anti-inflammatory medications. This will be assessed on a case by case basis by QI medical advisor.
* Drink more than 14 alcohol units/week.
* Smoke socially or on occasion more than 12.5 grams or 20 cigarettes/week
* Vegan or any dietary restrictions that prevent the consumption of study soups or follow a diet programme which requires fasting for multiple days.
* Are a registered blood donor and have donated a large quantity of blood within the last 16 weeks. Registered blood donors should abstain from blood donations for the duration of the study.
* Are unable to give written or verbal informed consent
* Unable to provide GP contact details.
* Are participating in another dietary intervention study nor given blood in another dietary study in the last 3 months.
* Are related to or living with any member of the study team or part of the management/supervisory structure of the Chief Investigator.
* Have symptoms of COVID-19, been asked to self-isolate, or have been diagnosed with COVID-19 in the last 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) after broccoli and courgette soup interventions | Week: 0, 12, 24 and 36.
  Comparison of fasting blood for HbA1c at baseline and after soup interventions

SECONDARY OUTCOMES:
Change in postprandial capillary glucose concentration | 3.5 hours
  Capillary glucose concentration will be measured by finger prick after administration of a glucose challenge using a standardized 75g glucose beverage (GlucosePro). Measurements will be taken -15, -10, -5, 15, 30, 45, 60, 90, 120, 150, 180, 210 min post glucose beverage at Week: 0, 12, 24 and 36.
Change in fasting plasma glucose (mmol/l) after broccoli and courgette soup interventions | Week: 0 to12 and 24 to 36.
  Comparison of fasting plasma glucose between baseline and at 12 weeks and washout (24 weeks) and 36 weeks.
Change in fasting plasma insulin (mmol/L) after broccoli and courgette soup interventions | Week: 0 to12 and 24 to 36.
  Comparison of fasting plasma insulin between baseline and at 12 weeks and washout (24 weeks) and 36 weeks.
Change in fasting serum fructosamine (µmol/L) after broccoli and courgette soup interventions | Week: 0 to12 and 24 to 36.
  Comparison of fasting serum fructosamine between baseline and at 12 weeks as well as washout (24 weeks) and 36 weeks.
Change in fasting serum cholesterol (mmol/L) after broccoli and courgette soup interventions | Week: 0 to12 and 24 to 36.
  Comparison of fasting serum cholesterol between baseline and at 12 weeks as well as washout (24 weeks) and 36 weeks.
Change in fasting serum triglycerides (mmol/L) after broccoli and courgette soup interventions | Week: 0 to12 and 24 to 36.
  Comparison of fasting serum triglycerides between baseline and at 12 weeks as well as washout (24 weeks) and 36 weeks.
Change in broccoli metabolites (glucosinolates, sulforaphane, and S-methyl cysteine sulfoxide) in 24 hour urine collection | Week: 0, 12, 24, and 36.
  Quantification of broccoli metabolite excretion into urine metabolites will be measured from 24-hour urine collections using targeted metabolite analysis of glucosinolates, sulforaphane, and S-methyl cysteine sulfoxide. These metabolites will be used to define relationships between dietary intake, broccoli metabolism and the biological outcomes
Treatment effects on whole blood gene expression from RNAseq | up to 36 weeks.
  The effect of soup consumption will be tested using edgeR and Limma to fit linear models to gene expression data. False discovery rate will be corrected using the Benjamin Hochberg procedure

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Kroon, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT05367024/Prot_SAP_000.pdf